CLINICAL TRIAL: NCT05378529
Title: A Multicenter, Cross-sectional Study to Characterize the Distribution of Lipoprotein(a) Levels Among Patients With Documented History of Atherosclerotic Cardiovascular Disease
Brief Title: A Cross-sectional Study of Lipoprotein(a) Levels in Patients With Documented History of Atherosclerotic Cardiovascular Disease (ASCVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20210057
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerotic Cardiovascular Disease; Lipoprotein(a)
MeSH Terms: conditions — Atherosclerosis | interventions — Apolipoproteins A; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with history of ASCVD (Other): Participants with history of ASCVD with known or unknown Lp(a) values.
  Interventions: Other: Lp(a) Screening

INTERVENTIONS:
Other: Lp(a) Screening — Participants will provide demographic information and have a blood draw for Lp(a) levels if they are unknown.

SUMMARY:
The purpose of this study is to characterize the distribution of lipoprotein(a) (Lp(a)) levels among participants with a history of ASCVD as defined by their medical history and is 2-fold:

* Evaluate the distribution of Lp(a) value in the overall participants with documented history of ASCVD
* Evaluate the distribution of Lp(a) value in participants with documented history of ASCVD by demographics and regions

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* History of ASCVD

Exclusion Criteria:

* Participants known to be currently receiving investigational drug in a clinical study
* Participants with a diagnosis of end-stage renal disease or requiring dialysis
* Participants who have received lipoprotein apheresis to reduce Lp(a) within 3 months prior to enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39480 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with elevated Lp(a) with documented history of ASCVD | Up to approximately 2 weeks

SECONDARY OUTCOMES:
Lp(a) Levels | Up to approximately 2 weeks
  Blood sampling will be performed in cases where Lp(a) values are not available at enrollment. In cases where Lp(a) values are available, data will be collected retrospectively.
Lp(a) Levels stratified by demographics and region | Up to approximately 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (735):
- United States (113):
  - Ascension Saint Vincents Birmingham, Birmingham, Alabama
  - Grandview Medical Center Affinity Cardiovascular Specialists, LLC, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Mobile Heart Specialists PC, Mobile, Alabama
  - Alaska Cardiovascular Research Foundation, Anchorage, Alaska
  - Care Access - Mesa, Mesa, Arizona
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Care Access - Berkeley, Berkeley, California
  - National Heart Institute, Beverly Hills, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - America Clinical Trials, Tarzana, California
  - Med Partners, Inc dba Premiere Medical Center, Inc, Toluca Lake, California
  - UCHealth Memorial Central, Colorado Springs, Colorado
  - Cardiology Associates of Fairfield County PC, Stamford, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Bay Area Cardiology, Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Cardiology Associates Research LLC, Daytona Beach, Florida
  - The Cardiac and Vascular Institute Research, Gainesville, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - Jellinger and Lerman MD PA dba The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - East Coast Institute for Research LLC at Northeast Florida Endocrine and Diabetes Research Associate, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - East Coast Institute for Research LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Advanced Research for Health Improvement, LLC, Naples, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Millennium Physician Group, LLC dba Charlotte Heart Group Research Center, Port Charlotte, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - Saint Johns Center for Clinical Research, Saint Augustine, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Care Access - Moss Bluff, Spring Hill, Florida
  - Care Access - Pebble Beach, Sun City, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Northeast Georgia Medical Center Wisteria Building, Cumming, Georgia
  - Northside Clinical Research, Johns Creek, Georgia
  - Care Access - Rome, Rome, Georgia
  - St Lukes Idaho Cardiology Associates, Meridian, Idaho
  - Northwest Heart Clinical Research LLC, Arlington Heights, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Saint Elizabeth Covington, Covington, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Louisiana Heart Center, Hammond, Louisiana
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - Monroe Research LLC, Monroe, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants LLC, Beltsville, Maryland
  - TidalHealth Peninsula Regional, Inc, Salisbury, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Arcturus Healthcare, Public Limited Company, Troy Internal Medicine Research Division, Troy, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Fairview Health Services, Saint Paul, Minnesota
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Bryan Heart, Lincoln, Nebraska
  - Palm Research Center Inc, Las Vegas, Nevada
  - Renown Institute for Heart and Vascular Health, Reno, Nevada
  - Saint Michaels Medical Center, Newark, New Jersey
  - New York Presbyterian Medical Group Hudson Valley Cardiology, Cortlandt Manor, New York
  - WMCHealth Heart and Vascular Institute Kingston Division of Cardiology, Kingston, New York
  - New York University Langone Health, New York, New York
  - Northwell Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Care Access - Bronx, The Bronx, New York
  - NY Family Docs, Woodhaven, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cone Health, Greensboro, North Carolina
  - Crossroads Clinical Research Inc, Mooresville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Rama Research LLC, Marion, Ohio
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Midlands Cardiology, Columbia, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Baylor Scott and White Heart and Vascular Hospital-Dallas, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Care Access - Georgetown, Georgetown, Texas
  - Baylor College of Medicine, Houston, Texas
  - Care Access - Katy, Katy, Texas
  - South Texas Cardiovascular Consultants, Kerrville, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Permian Research Foundation, Odessa, Texas
  - South Texas Cardiovascular Consultants PLLC, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Heart and Vascular Institute, Fairfax, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Bon Secours Cardiology, Midlothian, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Newport News, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Pulse Heart Institute, Puyallup, Washington
- Argentina (27):
  - Inst. de Inv. Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - CEDIC Centro de Investigacion Clinica, CABA, Buenos Aires
  - CIPREC - Centro de Investigacion y Prevencion Cardiovascular, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Consultorio Medico Dr Litvak Bruno, CABA, Buenos Aires
  - Centro de Especialidades Medicas - Cemedic, CABA, Buenos Aires
  - Centro Medico Dra LAURA MAFFEI e Investigacion clinica aplicada, CABA, Buenos Aires
  - Centro Medico Dra De Salvo, CABA, Buenos Aires
  - Consultorios Medicos Dr. Besada, CABA, Buenos Aires
  - Glenny Corp SA, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - ICBA - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Cuidad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Ciad - Consultorio Integral de Atencion al Diabetico, Morón, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - DIM Centros de Salud, Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clinicas de San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Clinica Privada del Prado, Córdoba, Córdoba Province
  - Instituto Latinoamericano de Investigaciones Medicas CIDIM-ILAIM, Córdoba, Córdoba Province
  - Instituto de Investigaciones Clinicas de Cordoba, Córdoba, Córdoba Province
  - Clinica Fusavim Privada SRL, Villa María, Córdoba Province
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Clinica Adventista Belgrano, Buenos Aires
  - Instituto Medico DAMIC, Córdoba
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Australia (22):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Advara HeartCare Wesley, Auchenflower, Queensland
  - Advara HeartCare Bundaberg, Bundaberg, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Dr Heart Pty Ltd, Woolloongabba, Queensland
  - Nightingale Research, Adelaide, South Australia
  - SA Heart, Ashford, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Advara HeartCare Berwick, Berwick, Victoria
  - Advara HeartCare Ringwood, Bundoora, Victoria
  - The Cardiologists Proprietary Limited, Epping, Victoria
  - Barwon Health Geelong Hospital, Geelong, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
  - Clinitrials, Murdoch, Western Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Krankenhaus der Barmherzigen Brueder Linz, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (14):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis - campus Aalst, Aalst
  - Ziekenhuisnetwerk Antwerpen site Cadix, Antwerp
  - Cliniques universitaires de Bruxelles Hopital Erasme, Brussels
  - Algemeen Ziekenhuis Sint Blasius, Dendermonde
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Algemeen Ziekenhuis Sint-Maarten, Mechelen
  - Sint-Trudo Ziekenhuis, Sint-Truiden
  - Algemeen Ziekenhuis Turnhout, Turnhout
- Brazil (39):
  - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Centro de Pesquisas em Diabetes e Doencas Endocrino Metabolicas, Fortaleza, Ceará
  - Hospital Universitario Walter, Vitória, Espírito Santo
  - Hospital Santa Izabel, Salvador, Estado de Bahia
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Salvador, Estado de Bahia
  - Associacao de Amparo a Saude Ensino e Pesquisa, Brasília, Federal District
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Universitario Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Eurolatino Pesquisas Medicas, Uberlândia, Minas Gerais
  - Quanta Diagnostico por Imagem, Curitiba, Paraná
  - Nucleo de Pesquisa Clinica, Curitiba, Paraná
  - Procape, Recife, Pernambuco
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital Sao Francisco da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Imv Pesquisa Cardiologica, Porto Alegre, Rio Grande do Sul
  - FZ Pesquisa e Servicos em Cardiologia LTDA, Porto Alegre, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - jmf Clinica do Coracao ltda, Aracaju, Sergipe
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - icm Instituto do Coração de Marilia, Marília, São Paulo
  - Clinicor Clinica Cardiologica Ltda, Ribeirão Preto, São Paulo
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto de Pesquisa em Endocrinologia Clinica IPEC, São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Fundacao Pro-Coracao, Rio de Janeiro
  - Centro Paulista de Investigacoes Clinicas Cepic, São Paulo
  - Instituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Bulgaria (13):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - Multiprofile Hospital for Active Treatment - Haskovo AD, Haskovo
  - Medical Center Medconsult Pleven OOD, Pleven
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - Medical Center Cardiomed 2020 EOOD, Sliven
  - Diagnostic-Consultative Center Ascendent OOD, Sofia
  - Multiprofile Hospital for Active Treatment National Hospital of Cardiology EAD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Kalimat EOOD, Sofia
  - Medical Centre Synexus Sofia EOOD, Sofia
  - Medical Center Orpheus OOD, Stara Zagora
  - Ambulatory for Individual Practice for Specialized Medical Care - Kardio EOOD, Varna
- Canada (14):
  - St Pauls Hospital, Vancouver, British Columbia
  - Discovery Clinical Services Ltd, Victoria, British Columbia
  - LMC Clinical Research Incorporated, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - LMC Clinical Research Incorporated Thornhill, Concord, Ontario
  - Hamilton Health Sciences Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - One Heart Care, Mississauga, Ontario
  - Oakville Cardiovascular Research, Oakville, Ontario
  - Ecogene-21 Research, Chicoutimi, Quebec
  - Institut de recherches cliniques de Montreal, Montreal, Quebec
  - Research Institute of McGill University Health Center - Glen Site, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - Clinique des Maladies Lipidiques de Quebec Incorporated, Québec, Quebec
- China (39):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital ,Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Huizhou Central Peoples Hospital, Huizhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Nanning Peoples Hospital, Nanning, Guangxi
  - Daqing Oilfield general Hospital, Daqing, Heilongjiang
  - Nanyang Second General Hospital, Nanyang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Second Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - Jilin Province Peoples Hospital, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Peoples Hospital of Liaoning Province, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Qingdao Fuwai Cardiovascular Hospital, Qingdao
  - Shanghai General Hospital, Shanghai
  - Shanghai Yangpu District Central Hospital（ Yangpu Hospital Affiliated to Tongji University）, Shanghai
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhejiang Hospital, Zhejiang
- Czechia (40):
  - Jessenia as, Nemocnice Beroun, Beroun
  - Hornicka nemocnice s poliklinikou spol sro, Bílina
  - Medicus Services sro, Brandýs nad Labem
  - MUDr Libor Nechvatal sro, Brno
  - Centrum pro zdravi sro, Brno
  - MUDr Karel Kameník sro, Brno
  - Kardiologicka ambulance Brno sro, Brno
  - Kardio Elbl sro, Brno
  - Edumed sro, Broumov
  - Ordinace pro choroby srdce sro, Chomutov
  - Nemocnice Ceske Budejovice as, České Budějovice
  - Dika centrum sro, Havirov - Mesto
  - CTC Hodonin sro, Cevni ambulance, Hodonín
  - Kardio Holesov sro, Holešov
  - MUDr Ladislava Harrerova, kardiologicka ordinace, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava po, Jihlava
  - Kardio Michal Cepelak sro, Klatovy IV
  - MUDr Zbynek Kosek, kardiologicka ambulance sro, Mladá Boleslav
  - PreventaMed sro, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Mestska nemocnice Ostrava, po, Ostrava - Moravska Ostrava
  - Pedicor Trial sro, Ostrava-Dubina
  - Nemocnice Pardubickeho kraje as, Pardubice
  - Fakultni nemocnice Plzen, Pilsen
  - Policska nemocnice sro, Polička
  - Ordinace pro choroby srdce a cev, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Pratia Prague sro, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Milan Kvapil sro, Prague
  - Interni a kardiologicka ordinace, Prague
  - Endokrinologie Cerny Most sro, Prague
  - Kardiologicke centrum MUDr Janky Skrobakove sro, Praha 5 - Smichov
  - Poliklinika Ravak Pribram, Pribram VIII
  - Kardio Vaclavik sro, Interni a kardiologicka ambulance, Přerov
  - Kardiologicka ambulance MUDr Ferkl, sro, Trutnov
  - Clinical Trials Service sro, Uherské Hradiště
  - Cardio Research sro, Zlín
  - Krajska nemocnice T Bati as, Zlín
- Denmark (16):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Sydvestjysk Sygehus, Esbjerg
  - Sanos Gandrup, Gandrup
  - Herlev Gentofte Hospital, Herlev
  - Sanos Clinic, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Holbaek Sygehus, Holbæk
  - Bispebjerg/Frederiksberg Hospitaler, København NV
  - Amager Hospital, København S
  - Odense University Hospital, Odense C
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Slagelse Sygehus, Slagelse
  - Svendborg Sygehus, Svendborg
  - Sanos Vejle, Vejle
  - Regionshospitalet Viborg, Viborg
- Estonia (5):
  - Innomedica, Tallinn
  - Center for Clinical and Basic Research Tallinn, Tallinn
  - Dr Arvo Rosenthal LLC, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Satucon Oy/Kuopion tyoterveys, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Suomen Terveystalo Oy, Turku
- France (20):
  - Centre Hospitalier Regional Universitaire de Besancon, Hopital Jean Minjoz, Besançon
  - Hospices Civils de Lyon Groupement Hospitalier Est, Hopital Louis Pradel, Bron
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Compiegne-Noyon, Compiègne
  - Centre Hospitalier Universitaire de Dijon - Hopital Francois Mitterrand, Dijon
  - Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Hopital de la Conception, Marseille
  - Hopital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Montpellier - Hopital Lapeyronie, Montpellier
  - Centre Hospitalier Universitaire de Nantes - Hopital Guillaume et Rene Laennec, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier Universitaire de Reims - Hopital Robert Debre, Reims
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Strasbourg - Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Polyclinique Vauban, Valenciennes
- Germany (27):
  - Universitaetsklinikum Aachen, Aachen
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Universitaetsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Klinische Forschung Berlin GbR, Berlin
  - Charite - Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Klinikum Links der Weser, Bremen
  - Universitaetsklinikum Koeln, Cologne
  - Diabetologische Gemeinschaftspraxis Dr Schaper und Dr Faulmann, Dresden
  - Universitaetsklinikum Dresden, Medizinische Klinik und Poliklinik III, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsmedizin Goettingen - Georg-August-Universitaet, Göttingen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Cardiologicum Hamburg GbR, Hamburg
  - B Braun Ambulantes Herzzentrum Kassel mvz GmbH, Kassel
  - Universitaetsklinikum Leipzig, Leipzig
  - Otto von Guericke Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitaetsklinikum Mannheim, Mannheim
  - Kardiologische Praxis Doktor Jens Taggeselle, Markkleeberg
  - Universitaetsklinikum Muenster, Münster
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Lipidambulanz der Universitaet Rostock, Rostock
  - Klinik am See - Ruedersdorf, Rüdersdorf
  - Hegau-Bodensee-Klinikum Singen, Singen
  - Forschungszentrum Ruhr, Witten
- Greece (13):
  - General Hospital of Athens Evaggelismos, Athens
  - Athens Naval Hospital, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - Laiko General Hospital, Athens
  - Alexandra Hospital, Athens
  - Attikon Hospital, Athens
  - Konstantopoulio - Agia Olga Hospital of Nea Ionia, Athens
  - Hygeia Hospital, Athens
  - Metropolitan Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Mitilini Vostanio, Mytilene
  - General Hospital of Thessaloniki Ahepa, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- Hungary (22):
  - Lausmed Kft, Baja
  - Dr Lakatos Ferenc Private Cardiology Practice, Békéscsaba
  - Budapesti Szent Ferenc Korhaz, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - High Tech Medical Kft, Budapest
  - Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet, Budapest
  - Del-budai Centrumkorhaz Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Semmelweis Egyetem Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Eszak-Pesti Centrum Korhaz - Honvedkorhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Kft, Encs
  - Pharma4 Trial Kft, Gyöngyös
  - BKS Research Kft, Hatvan
  - CRU Hungary Kft, Kistarcsa
  - Selye Janos Korhaz, Komárom
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Dr Nagy Laszlo Kardiologiai maganrendeles es SMO, Orosháza
  - Vita Verum Medical Bt, Székesfehérvár
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Belvarosi Egeszseghaz Kft, Zalaegerszeg
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Hjartamidstodin, Kopavogur, Iceland
- Italy (20):
  - Ospedali dell Ovest Vicentino, Arzignano
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Sant Anna e San Sebastiano, Caserta
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro
  - Azienda Ospedaliera Universitaria di Ferrara Arcispedale Sant Anna, Ferrara
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Maggiore della Carita, Novara
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale degli Infermi di Rivoli, Rivoli
  - Fondazione Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Policlinico Umberto I, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
  - Azienda Ospedaliera Universitaria Ospedale San Giovanni di Dio e Ruggi D Aragona, Salerno
  - Multimedica, Sesto San Giovanni (MI)
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (56):
  - Kasugai Municipal Hospital, Kasugai-shi, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - New Tokyo Heart Clinic, Matsudo-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu-shi, Fukuoka
  - Gifu Heart Center, Gifu, Gifu
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Hakodate Municipal Hospital, Hakodate-shi, Hokkaido
  - Tomakomai City Hospital, Tomakomai-shi, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa Medical University Hospital, Kahoku-gun, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Tenyoukai Chuo Clinic, Kagoshima, Kagoshima-ken
  - Fujisawa City Hospital, Fujisawa-shi, Kanagawa
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - Yokohama Sakae Kyosai Hospital Federation of National Public Service Personnel Mutual Association, Yokohama, Kanagawa
  - Chikamori Hospital, Kochi, Kochi
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - National University Corporation Tohoku University Tohoku University Hospital, Sendai, Miyagi
  - Sendai Cardiovascular Center, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Shinshu University Hospital, Matsumoto-shi, Nagano
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kawasaki Medical School Hospital, Kurashiki-shi, Okayama-ken
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Higashiosaka City Medical Center, Higashiosaka-shi, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Police Hospital, Osaka, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Saga-ken Medical Centre Koseikan, Saga, Saga-ken
  - Ageo Central General Hospital, Ageo-shi, Saitama
  - Kawaguchi Cardiovascular and Respiratory Hospital, Kawaguchi-shi, Saitama
  - Sanai Hospital, Saitama-shi, Saitama
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun, Shizuoka
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Minamino Cardiovascular Hospital, Hachioji-shi, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino-shi, Tokyo
  - Ome Medical Center, Ome-shi, Tokyo
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Seiyu Memorial Hospital, Wakayama, Wakayama
  - Tokuyama Central Hospital, Shunan-shi, Yamaguchi
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi
- Lithuania (6):
  - Klinikiniai sprendimai, Alytus
  - Klinikiniai sprendimai, Kaunas
  - Saules Seimos Medicinos Centras, Kaunas
  - Kardiologijos ir reabilitacijos klinika, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Vilnius University Hospital Santaros Clinic Public Institution, Vilnius
- Mexico (5):
  - Eukarya PharmaSite S.C., Monterrey, Nuevo León
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada SC, Culiacán, Sinaloa
  - Fundacion Cardiovascular de Aguascalientes AC, Aguascalientes
  - Scientia Investigacion Clinica SC, Chihuahua City
  - Procliniq Investigación Clínica Sa de Cv, Mexico City
- Netherlands (30):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Bravis Ziekenhuis, Bergen op Zoom
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Spaarne Gasthuis, locatie Haarlem Zuid, Hoofddorp
  - Dijklander Ziekenhuis Hoorn, Hoorn
  - Leids Universitair Medisch Centrum, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - D and A Research and Genetics, Sneek
  - Haaglanden MC, The Hague
  - Haga Ziekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
- Norway (3):
  - Oslo Universitetssykehus HF Aker sykehus, Oslo
  - Oslo Universitetssykehus HF, Aker sykehus, Oslo
  - Skedsmo Medisinske senter, Skedsmokorset
- Poland (20):
  - American Heart of Poland Spolka Akcyjna, Bełchatów
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Bielsko-Biala
  - American Heart of Poland Spolka Akcyjna, Chrzanów
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Dąbrowa Górnicza
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ Medica Jerzy Cygler, Giżycko
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Kędzierzyn-Koźle
  - Jaroslaw Ciosek Rajtar-Medica Centrum Medyczne, Krakow
  - Wojewodzki Specjalistyczny Szpital im dr Wladyslawa Bieganskiego w Lodzi, Lodz
  - CenterMed Spzoo Centermed Lublin, Lublin
  - Clinical Best Solutions Sp zoo Spolka Komandytowa Gabinet Lekarski, Lublin
  - NZOZ Twoja Przychodnia Spzoo, Lublin
  - Uniwersyteckie Centrum Stomatologii I Medycyny Specjalistycznej Spolka z ograniczona odpowiedzialnos, Poznan
  - American heart of poland spolka skcyjna polsko amerykanskie kliniki serca, Poznan
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Sztum
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Tychy
  - Szpital Grochowski imienia Doktora medycyny Rafala Masztaka Spzoo, Warsaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Samodzielny Publiczny Szpital Wojewodzki im Papieza Jana Pawla II w Zamosciu, Zamość
  - American Heart of Poland Spolka Akcyjna, Zgierz
- Portugal (10):
  - Hospital Professor Doutor Fernando Fonseca, EPE, Amadora
  - Centro Hospitalar do Baixo Vouga, EPE - Hospital Infante Dom Pedro, Aveiro
  - Hospital de Braga, EPE, Braga
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Centro Hospitalar e Universitario de Coimbra EPE, Coimbra
  - Hospital da Senhora da Oliveira Guimaraes, EPE, Guimarães
  - Unidade Local de Saude de Matosinhos - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar de Entre o Douro e Vouga, EPE - Unidade de Sao Sebastiao, Santa Maria da Feira
  - Centro Hospitalar de Setubal EPE Hospital de Sao Bernardo, Setúbal
  - Centro Hospitalar de Vila Nova de Gaia/Espinho EPE, Vila Nova de Gaia
- Romania (10):
  - cmi Cardiologie - Dr Mercea Corina Delia, Baia Mare
  - Spitalul Universitar de Urgenta Militar Central Dr Carol Davila, Bucharest
  - Spitalul Clinic Universitar de Urgenta Elias, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Matcord Biomedica Buzau, Buzău
  - SC Sal Med SRL, Piteşti
  - Cardio Med Medical Center Targu Mures, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Clinica Medicalis Timisoara, Timișoara
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Slovakia (23):
  - Alian, sro, Bardejov
  - Remedium, sro, Bardejov
  - Narodny ustav srdcovych a cievnych chorob, as, Bratislava
  - Kardiovita sro, Bratislava
  - Nemocnica s poliklinikou Brezno, no, Brezno
  - La-Ro Cor sro, Handlová
  - Intergal, sro, Kláštor pod Znievom
  - Medical group Kosice sro, Košice
  - Zarmed, sro, Košice
  - Cardio D and R, sro Kosice, Košice
  - Kardio 1 sro, Lučenec
  - Medi M and M sro, Moldava nad Bodvou
  - Oralek, sro, Námestovo
  - Kardiocentrum Nitra sro, Nitra
  - Kardiomed NZ, sro, Nové Zámky
  - Benimed sro, Piešťany
  - Medikard, sro, Prešov
  - Medispol, sro, Prešov
  - Medilex sro, Rimavská Sobota
  - Tatratrial sro, Rožňava
  - Interna SK, sro, Svidník
  - Areteus sro, Trebišov
  - CardiOr, sro, Trenčín
- South Korea (15):
  - Dong-A University Hospital, Busan
  - Keimyung University, Dongsan Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (22):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario de Leon, León, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital de Sant Joan Despi Moises Broggi, Sant Joan Despí, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia, Valencia
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (8):
  - Ladulaas Kliniska Studier, Borås
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Clemenstorgets Hjartmottagning, Lund
  - PharmaSite Malmo, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (5):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Istituto Cardiocentro Ticino, Lugano
  - Kantonsspital St Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- Taiwan (10):
  - Hualien Tzu Chi Hospital, Hualien City, Hualien
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Mackay Memorial Hospital Tamsui Branch, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (20):
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Adana
  - Afyonkarahisar Saglik Bilimleri Universitesi Hastanesi, Afyonkarahisar
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Adnan Menderes Universitesi Medical Faculty, Aydin
  - Koc Universitesi Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bagcilar Egitim ve Arastirma Hastanesi, Istanbul
  - Dr Siyami Ersek Gogus Kalp ve Damar Cerrahisi Egitim ve Arastirma Hastanesi, Istanbul
  - Kartal Kosuyolu Yuksek Ihtisas Egitim ve Arastirma Hastanesi, Istanbul
  - Tepecik Egitim ve Arastirma Hastanesi, Izmir
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi, Izmir
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
  - Sitki Kocman Universitesi, Muğla
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
  - Van Yuzuncu Yil Universitesi Dursun Odabas Tip Merkezi, Van
- United Kingdom (32):
  - Aberdeen Royal Infirmary, Aberdeen
  - Ormeau Clinical Trials Ltd, Belfast
  - Russell Hall Hospital, Birmingham
  - NIHR Patient Recruitment Centre Blackpool, Blackpool
  - NIHR Patient Recruitment Centre Bradford, Bradford
  - West Walk Surgery, Bristol
  - St Richards Hospital, Chichester
  - Craigavon Area Hospital, Craigavon
  - Panthera Biopartners - London, Enfield
  - NIHR Patient Recruitment Centre Exeter, Exeter
  - Panthera Biopartners - Glasgow, Glasgow
  - Harefield Hospital, Harefield
  - Wycombe General Hospital, High Wycombe
  - Hull Royal Infirmary, Hull
  - Highlands Clinical Research Facility, Raigmore Hospital, Inverness
  - NIHR Patient Recruitment Centre Leicester, Leicester
  - Lincoln County Hospital, Lincoln
  - Royal Liverpool University Hospital, Liverpool
  - Queen Mary University of London, London
  - Hammersmith Hospital, London
  - Wythenshawe Hospital, Manchester
  - NIHR Patient Recruitment Centre Newcastle, Newcastle
  - Nottingham City Hospital, Nottingham
  - University Hospital Llandough, Penarth
  - The Adam Practice, Poole
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Rochdale, Rochdale
  - Ashfield Primary Care Centre, Sandbach
  - Lister Hospital, Stevenage
  - Princess Royal Hospital, Telford
  - Rowden Surgery, Wilts
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com